CLINICAL TRIAL: NCT01561742
Title: Minocycline Augmentation in Early-Course Schizophrenia
Brief Title: Minocycline Augmentation in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Mujeeb Shad, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-11-0201
Record Dates: First submitted 2012-03-14; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia
Keywords: minocycline, augmentation, schizophrenia
MeSH Terms: conditions — Schizophrenia; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental)
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — Minocycline will be given orally at 200 mg a day for 4 months
  Other Names: Minocin
  Arms: Minocycline
Drug: Placebo — EquivalentPlacebo will be given
  Arms: Placebo

SUMMARY:
This study aims to examine the efficacy of minocycline augmentation in a sample of moderately ill outpatients with early-course schizophrenia on their chlorpromazine-equivalent doses of second-generation antipsychotic medications. The investigators hypothesize that as compared to placebo a 2-month treatment with minocycline in 120 volunteers with early-course schizophrenia will result in a more significant improvement in psychopathology (primary outcome) and cognitive symptoms (secondary outcome). In addition, cytokine plasma levels will be used as another secondary outcome measure to see if treatment-induced changes in total PANSS score are associated with changes in cytokine levels.

DETAILED DESCRIPTION:
Minocycline, which is a second-generation tetracycline, has been found to inhibit Nitric Oxide Synthase (NOS) and inflammatory cytokines. These are some of the primary mechanisms that have been proposed to explain its neuroprotective and neuroplastic effects in several animal and human models of neurological and psychiatric diseases, including Parkinson's disease and schizophrenia. There are only three clinical trials with minocycline in schizophrenia subjects. A more definitive clinical trial in a larger sample with optimized and cost-effective design using a comprehensive cognitive battery and a global assessment of schizophrenia symptom domains is necessary to examine the efficacy of minocycline. If minocycline improves psychopathology and potentially other symptoms (including cognitive function) for schizophrenia, the treatment could be easily implemented in the existing treatment delivery system at relatively low cost and have the potential for making a significant public health impact. The investigators plan to recruit 120 individuals with early course schizophrenia who are currently on second-generation antipsychotic (SGA) medications and are experiencing persistent symptoms in at least the moderate range. In an effort to limit placebo response, which is notoriously high in psychiatric population, the investigators are using an adaptive design. Since, there is growing evidence to support the inflammatory hypothesis of schizophrenia, the investigators will also explore whether cytokine levels mediate the response from minocycline treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18-35 years
2. Males & females
3. Current DSM-IV diagnosis of schizophrenia or schizoaffective disorder confirmed by the Mini-International Neuropsychiatric Interview (M.I.N.I.) conducted by a trained psychiatrist.
4. Treatment with a stable dose of second generation antipsychotic medication for at least 1 months prior to study entry 200-600 mg/day chlorpromazine equivalent doses);
5. Evidence of stable symptomatology for 12 weeks as evidenced by no hospitalizations for schizophrenia, no increase in level of psychiatric care due to worsening of symptoms, no ER use for symptoms of schizophrenia and no significant changes to antipsychotic medication or dose (>25%) in the past 12 weeks.
6. Baseline total score between 40 and 65 on the Brief Psychiatric Rating Scale (BPRS);
7. Raw score of 12 or higher on the Wechsler Test of Adult Reading (WTAR) (estimates premorbid IQ).
8. Able to comprehend the procedure and aims of the study to provide informed consent

Exclusion Criteria:

1. Acute, unstable, significant or untreated medical illness beside schizophrenia;
2. Pregnant or breast-feeding females;
3. History of substance abuse or dependence in the past 3 months.
4. Known contraindication to minocycline treatment.
5. Treatment with minocycline or Beta-lactam antibiotics in the preceding half year before study entry.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-induced change in total score on Positive and Negative Syndrome Scale (PANSS) | Baseline, week 8, and week 16 of the study
  PANSS total score will be used to examine treatment-induced change in psychaopthology. The PANSS is a 30-item rating scale used to assess symptoms of psychopathology. We will use the total PANSS score as the primary outcome measure which reflects total level of psychopathology including the positive and negative symptoms as well as general psychopathology.This measure will be administered at baseline, week 8 and week 16 of the study to assess if minocyline treatment results in a significant reduction in PANSS total score as opposed to placebo.

SECONDARY OUTCOMES:
Treatment-induced change in MATRICS Cognitive Consensus Battery (MCCB) | Baseline and week 16 of the study
  Average total score on MCCB will be used to examine treatment-induced change in cognitive function. MCCB (Nuechterlein et al., 2008) will be admisnitered at the baseline an week 16 of the study. The MCCB assesses 7 domains of cognitive functioning known to be impaired for individuals with schizophrenia. A summary score averaging across domains is generated as a global measure of cognitive functioning.
Treatment-induced changes in plasma level of cytokines | Baseline and week 16 of the study
  Cytokine levels will assessed at baseline and week 16 of the study to examine treatment-induced changes in neuroinflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Mujeeb U Shad, MD, MSCS, Principal Investigator — UT Health Sciences Center at Houston
Locations (1):
- Harris County Psychiatric Center, Houston, Texas, United States